CLINICAL TRIAL: NCT05195333
Title: Comparison of Home Exercises and Home Exercise Pogram Taught by Physiotherapist in Women With Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Principle Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Merveymz.
Record Dates: First submitted 2021-12-30; First posted 2022-01-18 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; home exercise; physiotherapist
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know which group to belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First group (Experimental): The exercise program prepared for the 1st group gestational diabetes will be explained to the pregnant women by the physiotherapist and the exercises will be taught to the patient. You will be asked to do these exercises as home exercise with 10 repetitions 3 days a week, until the 34th week of pregnancy.
  Interventions: Other: The exercise program
- Second group (Experimental): The same exercise program will be given to the participants only as a brochure and they will be asked to do 10 repetitions at home, 3 days a week, until the 34th week of pregnancy
  Interventions: Other: The exercise program
- Third group (No Intervention): The participants will not be given any exercise program, they will be asked to continue their routine care.

INTERVENTIONS:
Other: The exercise program — The exercise program prepared for the 1st group gestational diabetes will be explained to the pregnant women by the physiotherapist and the exercises will be taught to the patient.
  Arms: First group
Other: The exercise program — The same exercise program will be given to the participants only as a brochure and they will be asked to do 10 repetitions at home, 3 days a week, until the 34th week of pregnancy.
  Arms: Second group

SUMMARY:
Participants will be randomized and divided into 3 groups. The exercise program prepared for the 1st group gestational diabetes will be explained to the pregnant women by the physiotherapist and the exercises will be taught to the patient. They do these exercises as home exercise with 10 repetitions 3 days a week, until the 34th week of pregnancy. In the second group, the same exercise program will be given to the participants only as a brochure and they will be asked to do 10 repetitions at home, 3 days a week, until the 34th week of pregnancy. In the 3rd group, the participants will not be given any exercise program, they will be asked to continue their routine care.

DETAILED DESCRIPTION:
45 pregnant women who applied to Çamlıca Medipol Hospital Gynecology and Obstetrics and were diagnosed with gestational diabetes will be included in the study. Being between the ages of 20-40, pregnancy of 26-30 weeks, being diagnosed with gestational diabetes as a result of oral glucose tolerance test, BMI>45 kg/m2, being physically inactive are inclusion criteria. Exclusion criteria are being younger than 18 years of age, having a history of Type 1 or Type 2 diabetes, having undergone bariatric surgery, using drugs that cause weight gain, and contraindications that prevent exercise. Participants will be randomized and divided into 3 groups. The exercise program prepared for the 1st group gestational diabetes will be explained to the pregnant women by the physiotherapist and the exercises will be taught to the patient. They do these exercises as home exercise with 10 repetitions 3 days a week, until the 34th week of pregnancy. In the second group, the same exercise program will be given to the participants only as a brochure and they will be asked to do 10 repetitions at home, 3 days a week, until the 34th week of pregnancy. In the 3rd group, the participants will not be given any exercise program, they will be asked to continue their routine care. Participants' fasting glucose and HbA1c values, anthropometric measurements, physical activity levels with the "pregnancy physical activity questionnaire (GFAA) and their quality of life with the World Health Organization Quality of Life Scale Short Form will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-40 years old
* 26-30. week of pregnancy
* Diagnosis of gestational diabetes as a result of an oral glucose tolerance test
* BMI>45 kg/m2
* Being physically inactive

Exclusion Criteria:

* Being under the age of 18
* History of Type 1 or Type 2 diabetes
* Have had bariatric surgery
* Use of drugs that cause weight gain
* Contraindications preventing exercise

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 45 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy physical activity questionnaire for physical activity level measurement | 5 minutes
  It is a questionnaire that asks pregnant women to report their usual physical activities during the last month and questions the time spent with a total of 32 activities under the subheadings of housework/care activities, professional activities, sports/exercise.
HbA1c measurement | 10 minutes
  HbA1c values of the participants will be done in Medipol University laboratory.
Fasting glucose measurements | 10 minutes
  Fasting glucose values of the participants will be done in Medipol University laboratory.
World Health Organization Quality of life Short Form for measurement of quality of life | 5 minutes
  The scale measures physical, mental, social and environmental well-being and consists of 26 questions.

SECONDARY OUTCOMES:
Weight measurement | 2 minutes
  Weight in kilogram will be measured with weighing machine
Height measurement | 2 minutes
  Height in meters will be measured with tape measure
Body mass index (BMI) measurement | 2 minutes
  Weight and height will be combined to report BMI in kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will publish an article about the results of the study and share it with other researchers.

REFERENCES:
- [Result] Downs DS, Dinallo JM, Birch LL, Paul IM, Ulbrecht JS. Randomized Face-to-Face vs. Home Exercise Interventions in Pregnant Women with Gestational Diabetes. Psychol Sport Exerc. 2017 May;30:73-81. doi: 10.1016/j.psychsport.2017.02.003. Epub 2017 Feb 20. PMID 28428728
- [Derived] Menek MY, Kaya AK. Comparison of home exercise under supervision and self home exercise in pregnant women with gestational diabetes: randomized controlled trial. Arch Gynecol Obstet. 2024 Mar;309(3):1075-1082. doi: 10.1007/s00404-023-07339-4. Epub 2024 Jan 6. PMID 38184491
- See also: Randomized Face-to-Face vs. Home Exercise Interventions in Pregnant Women with Gestational Diabetes — https://pubmed.ncbi.nlm.nih.gov/28428728/